CLINICAL TRIAL: NCT01737008
Title: Phase I Trial of Dacomitinib Concomitant With Radiotherapy With and Without Cisplatin in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Dacomitinib Plus Radiotherapy, With and Without Cisplatin in Patients With Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XDC-001
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and neck; Squamous cell carcinoma; Phase 1; Dacomitinib; Radiation; Radiotherapy; Chemotherapy; Chemoradiation; Chemoradiotherapy; Cisplatin; Pharmacokinetics; Maximum tolerated dose; Safety; Human epidermal growth factor receptor; Previously Untreated; Local or Locally Advanced
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — dacomitinib; Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dacomitinib with Radiotherapy (Experimental): Dacomitinib, 15mg to 45mg orally, once daily. Radiotherapy, once daily (Monday to Friday) over six weeks.One day on weeks 2 to 6 the participants will receive treatment twice daily (bid).
  Interventions: Drug: dacomitinib; Radiation: Radiotherapy
- Dacomitinib and Chemoradiotherapy (Experimental): Dacomitinib: 15mg to 45mg orally, once daily. Radiotherapy: Once daily (Monday to Friday) over seven weeks. Twice daily (bid) treatments may be introduced to compensate for treatment days missed due to statutory holidays, or machine maintenance. Cisplatin: 100mg/m2 intravenously; weeks 1, 4, and 7.
  Interventions: Drug: dacomitinib; Radiation: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: dacomitinib — Tablets are administered orally or through a G-Tube, and can be taken with or without food.
  Other Names: PF-00299804
Radiation: Radiotherapy — Intensity modulated radiation therapy (IMRT) delivered using 4 or 6 MV photons. Patients will receive either the standard dose fractionation radiotherapy or accelerated fractionation radiotherapy.
Drug: Cisplatin — If selected for this arm, cisplatin will be administered intravenously every three weeks after receiving premedications.
  Other Names: cisplatinum
  Arms: Dacomitinib and Chemoradiotherapy

SUMMARY:
This is a phase 1 study of the drug dacomitinib with radiotherapy, with or without chemotherapy, in patients with advanced squamous cell carcinoma of the head and neck (SCCHN).

Dacomitinib is an oral drug, which is found to be active in SCCHN patients, blocks a receptor called the epidermal growth factor receptor (EGFR). By blocking signals for cancer cells to grow, it is believed to stop or slow the growth of tumor cells.

The dose escalation phase will find the best dose as well as determine the safety of dacomitinib when given with radiotherapy and with or without chemotherapy.The dose expansion phase will further test the best dose determined in the dose escalation phase for response rate.

DETAILED DESCRIPTION:
This is a phase 1 study of the investigational drug, dacomitinib, with radiotherapy and with or without chemotherapy in patients with advanced squamous cell carcinoma of the head and neck (SCCHN).

There are proteins found on the surface of cells called receptors that receive signals and send signals to the cell to grow or to die. Dacomitinib is an oral drug that blocks a receptor called the epidermal growth factor receptor (EGFR) which is found to be too active in SCCHN patients. By blocking the signals for the cancer cells to grow, it is believed to stop or slow the growth of tumor cells. The treatment of SCCHN usually includes chemotherapy and radiation.

The primary objectives of this study will have two phases: a dose escalation phase and a dose expansion phase. The dose escalation phase will find the best dose as well as determine the safety of dacomitinib when given with radiotherapy and with or without chemotherapy.The dose expansion phase will further test the best dose determined in the dose escalation phase for safety and response rate.

The secondary objectives are to evaluate the pharmacokinetic properties of the combination therapies, and to provide preliminary survival data.

ELIGIBILITY:
Inclusion Criteria:

* Signed voluntary informed consent provided.
* Patient willing and able to comply with visits, treatment plan, pharmacokinetics, laboratory tests, other study procedures.
* Escalation: Arm A: patients with local/locally advanced confirmed SCCHN; candidates for radical radiotherapy. Arm B: previously untreated patients, with locally advanced, confirmed SCCHN; candidates for radical concurrent cisplatin-based chemoradiation.
* Expansion: previously untreated patients, with locally advanced, confirmed SCCHN; HPV-negative candidates for radical concurrent cisplatin-based chemoradiation.Note: Those with primary tumors of head and neck in nasopharynx, skin, or unknown are excluded.
* Prior treatment of current neoplasm not allowed; must not have received any anti-neoplastic treatment within 2 years.
* Treatment-related toxicity must have recovered to CTCAE Grade 1 (v.4.0) or baseline, except toxicities not considered a risk. Chronic dysphagia, xerostomia or other effect resulting from prior surgery will not be considered exclusion criterion.
* ECOG performance status 0-1.
* Patient must have adequate organ function determined by: Creatinine clearance of ≥ 50 mL/min using formula: Creatinine clearance=[(140-age) x wt (kg) x Constant]/creatinine (µmol/L) [Constant = 1.23 for men; 1.04 for women]. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Leukocytes > 3.0 x 109/L; Hemoglobin > 80 g/L (or > 8 g/dL); Platelets ≥ 100 x 109/L. Total bilirubin ≤ ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN. 12-Lead electrocardiogram (ECG) with normal tracing, or clinically non-significant changes. QTc interval < 480 msec, without history of Torsades de Pointes or other QTc abnormality.

Exclusion Criteria:

* Enrollment in another clinical trial.
* Prior trial drug use within 30 days or 5 half-lives preceding first dose of study medication.
* Prior treatment with agents targeted to epidermal growth factor receptor
* Requirement for drugs highly dependent on CYP2D6 for metabolism - dacomitinib is a potent CYP2D6 inhibitor [See Appendix B and C].
* Patients taking drugs causing risk for Torsades de Pointes
* Any acute/chronic medical, psychiatric, laboratory abnormality that investigator finds could increase risks of participation, trial drug administration or could interfere with trial results. Including: History of interstitial lung disease; uncontrolled hypertension, unstable angina, myocardial infarction, symptomatic congestive heart failure within a year, cardiac arrhythmia, diagnosed/suspected congenital long QT syndrome; cardiovascular or vascular disease with anti arrhythmic therapy and/or major changes to medical care within 6 months; active bacterial, fungal or viral infection including hepatitis B or C, and human immunodeficiency virus. Testing not required for patients with no symptoms of infection. History of bleeding disorder, or concurrent medications the investigator finds to potentially lead to unacceptable coagulation function, including: congenital bleeding disorders; acquired bleeding disorder within one year; Other serious uncontrolled medical disorder or active infection that investigator determines may impair ability to receive study treatment. Dementia or altered mental status that limits ability to obtain informed consent and compliance with requirements of protocol.
* Breastfeeding/pregnancy. Females with reproductive potential [any female who had menarche and who has not had successful surgical sterilization/is not postmenopausal (defined as amenorrhea >12 consecutive months/women on hormone replacement therapy with serum follicle stimulating hormone level >35 mL.U/mL)] require negative pregnancy test within 72 hours of treatment.
* Patients of reproductive potential/partners must agree to effective contraception while receiving trial treatment and for 3 months after. Effective contraception will be judgment of principal investigator or designate.
* Inability or lack of willingness to comply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (in mg) of Dacomitinib | 1 year
To preliminarily evaluate the response rate of the combination of Dacomitinib, Cisplatin and Radiation | 1 year

SECONDARY OUTCOMES:
Levels of Dacomitinib in the Blood (Pharmacokinetics) in Combination with Cisplatin and Radiation | Days 8, 22 and 43 (+2 day window) after initial dose
Disease free survival, overall survival and locoregional and distant metastasis free survival | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, M.D., Principal Investigator — Princess Margaret Cancer Centre/University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chiu JW, Chan K, Chen EX, Siu LL, Abdul Razak AR. Pharmacokinetic assessment of dacomitinib (pan-HER tyrosine kinase inhibitor) in patients with locally advanced head and neck squamous cell carcinoma (LA SCCHN) following administration through a gastrostomy feeding tube (GT). Invest New Drugs. 2015 Aug;33(4):895-900. doi: 10.1007/s10637-015-0245-3. Epub 2015 May 5. PMID 25937431